CLINICAL TRIAL: NCT06884943
Title: Randomized Trial of AI-Enhanced Maintenance Training With Visual-Acoustic Biofeedback
Brief Title: Generalization With AI Navigation Using StaRt
Acronym: GAINS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Syracuse University (Other); Montclair State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRESULTS GAINS; 2R01DC017476 (NIH)
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-03

CONDITIONS: Speech Sound Disorder
Keywords: speech; articulation
MeSH Terms: conditions — Speech Sound Disorder; Speech | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants who meet criteria for inclusion in the GAINS follow-up study will be categorized into low and high severity groups and will be randomized with stratification by severity to the TAU and TAU+AI conditions. Participants will then complete 6 weeks in their randomly assigned condition.
Who Masked: Outcomes Assessor
Masking Description: All perceptual ratings will be obtained from blinded, naive listeners recruited through online crowdsourcing. Following protocols refined in previous published research, binary rating responses will be aggregated over at least 9 unique listeners per token.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-guided maintenance training with visual-acoustic biofeedback (Experimental): Participants will receive visual-acoustic biofeedback treatment from a clinician in a private, password-protected WebRTC room.
  Interventions: Behavioral: AI-guided maintenance training with visual-acoustic biofeedback; Behavioral: Treatment as Usual (TAU)
- Treatment as usual [TAU] (Active Comparator): Regular community-based care.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: AI-guided maintenance training with visual-acoustic biofeedback — Participants will complete AI-guided practice in the home setting in which they will interact with a web interface of the staRt web-based software for speech practice. The staRt software will present words to practice and show a real-time visual display of the acoustic signal of speech (biofeedback). On select trials, feedback will be provided by a classifier for children's "r" sounds, PERCEPT. Research assistants will join sessions to facilitate but will not provide direct clinical guidance to participants.
  Arms: AI-guided maintenance training with visual-acoustic biofeedback
Behavioral: Treatment as Usual (TAU) — Participants will return to their regular community-based care. This may consist of treatment in the school setting or by a private SLP; participants who were not previously receiving treatment may return to a no-treatment condition. Data will be collected from parents/guardians to determine the frequency of treatment, if any, received during this phase.

SUMMARY:
Speech Sound Disorder (SSD) affects a significant portion of school-aged children, leading to social and emotional challenges that can persist into adolescence and adulthood. The number of productions necessary for a remediated speech sound to generalize to connected speech is challenging to achieve in practice, leading clinicians to call for accessible, reliable resources allowing children to continue therapy outside of direct clinical interactions. Artificial intelligence (AI) tools hold promise as a means to extend direct service delivery in speech-language pathology, but research investigating the topic has been limited. This study (Generalization with AI Navigation using staRt, or GAINS) will measure the effects of a course of AI-mediated home practice intended to promote generalization of gains made through biofeedback treatment in a related study, Visual-acoustic Intervention with Service Delivery In-person and Via Telepractice Trial (VISIT; NCT06517225).

DETAILED DESCRIPTION:
This study will measure the effects of AI-guided home practice as a follow-up to participation in a study of technology-enhanced treatment for speech sound disorder affecting the American English "r" sound. Participants will sign a single consent form that covers their participation in the original VISIT study (in which they are randomized to receive biofeedback treatment in person or via telepractice) and and the follow-up GAINS study (in which participants are randomized to a follow-up period of treatment as usual [TAU] or treatment as usual plus an AI-guided maintenance program with biofeedback [TAU+AI]).We will measure production accuracy at the start and end of GAINS to test our working hypothesis that children/adolescents with speech sound disorder will show higher accuracy in /r/ production after six weeks of TAU+AI than six weeks of TAU alone. All GAINS treatment sessions will be carried out in the home setting using online tools. Pre and post treatment evaluations will be carried out in the laboratory setting.

ELIGIBILITY:
Inclusion Criteria:

* • Must be between 9;0 and 17;11 (years;months) old at the time of enrollment.

  * Must speak English as the dominant or equally dominant language
  * Must have begun learning English by age 3, per parent report.
  * Must hear a rhotic dialect of English from at least one speaker in the home if the home language is English.
  * Must pass a pure-tone hearing screening.
  * Must pass a brief examination of oral structure and function.
  * Must demonstrate age-appropriate receptive and expressive language abilities on the Clinical Evaluation of Language Fundamentals-5 (CELF-5).
  * Must have access to a laptop or desktop computer for study sessions.
  * Must have home wifi sufficient to support video calls in the event of randomization to the telepractice condition.
  * Must have completed participation in the VISIT randomized controlled trial.
  * Must score at least 60% correct in at least one treatment session during the related previous study, VISIT.

Exclusion Criteria:

* • Must not exhibit voice or fluency disorder of a severity judged likely to interfere with the ability to participate in study activities.

  * Must not currently have orthodontia that crosses the palate and cannot be removed.
  * Must not have history of permanent hearing loss.
  * Must not have an existing diagnosis of developmental disability such as cerebral palsy or Down Syndrome.
  * Must not have history of major brain injury, surgery, or stroke in the past year.
  * Must not have epilepsy with active seizure incidents with in the past 6 months.
  * Must not show clinically significant signs of apraxia of speech or dysarthria.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
1. Percentage of "Correct" Ratings by Blinded Untrained Listeners for /r/ Sounds Produced in Word Probes | Immediately before the initiation of GAINS participation and again after the end of GAINS participation (6 weeks later)
  To assess generalization of treatment gains to untreated words, participants will be assessed with standard probes (30 words [considered the primary target], 20 syllables, and 10 sentences containing /r/ in various phonetic contexts). Stimuli in each probe will be presented individually in randomized order with blocking by stimulus type (word, syllable, sentence). Individual words will be isolated from the audio record of each word probe and presented in randomized order for binary rating (correct/incorrect) by 9 untrained listeners who are blind to treatment condition and time point, but will see the written representation of each target word. We will use the proportion of "correct" ratings for each token as our primary measure of perceptually rated accuracy.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Montclair State University, Bloomfield, New Jersey
  - Syracuse University, Syracuse, New York

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, Analytic Code

REFERENCES:
- [Background] Ochs LC, Leece MC, Preston JL, McAllister T, Hitchcock ER. Traditional and Visual-Acoustic Biofeedback Treatment via Telepractice for Residual Speech Sound Disorders Affecting /ɹ/: Pilot study. Perspect ASHA Spec Interest Groups. 2023 Dec;8(6):1533-1553. doi: 10.1044/2023_persp-23-00120. Epub 2023 Nov 8. PMID 38764857
- [Background] Peterson L, Savarese C, Campbell T, Ma Z, Simpson KO, McAllister T. Telepractice Treatment of Residual Rhotic Errors Using App-Based Biofeedback: A Pilot Study. Lang Speech Hear Serv Sch. 2022 Apr 11;53(2):256-274. doi: 10.1044/2021_LSHSS-21-00084. Epub 2022 Jan 20. PMID 35050705
- [Background] Byun TM, Hitchcock ER. Investigating the use of traditional and spectral biofeedback approaches to intervention for /r/ misarticulation. Am J Speech Lang Pathol. 2012 Aug;21(3):207-21. doi: 10.1044/1058-0360(2012/11-0083). Epub 2012 Mar 21. PMID 22442281
- [Background] Byun TM, Hitchcock ER, Swartz MT. Retroflex versus bunched in treatment for rhotic misarticulation: evidence from ultrasound biofeedback intervention. J Speech Lang Hear Res. 2014 Dec;57(6):2116-30. doi: 10.1044/2014_JSLHR-S-14-0034. PMID 25088034
- [Background] McAllister Byun T, Halpin PF, Szeredi D. Online crowdsourcing for efficient rating of speech: a validation study. J Commun Disord. 2015 Jan-Feb;53:70-83. doi: 10.1016/j.jcomdis.2014.11.003. Epub 2014 Dec 15. PMID 25578293
- [Background] McAllister Byun T, Campbell H. Differential Effects of Visual-Acoustic Biofeedback Intervention for Residual Speech Errors. Front Hum Neurosci. 2016 Nov 11;10:567. doi: 10.3389/fnhum.2016.00567. eCollection 2016. PMID 27891084
- [Background] McAllister Byun T. Efficacy of Visual-Acoustic Biofeedback Intervention for Residual Rhotic Errors: A Single-Subject Randomization Study. J Speech Lang Hear Res. 2017 May 24;60(5):1175-1193. doi: 10.1044/2016_JSLHR-S-16-0038. PMID 28389677
- [Background] Hitchcock ER, Byun TM. Enhancing generalisation in biofeedback intervention using the challenge point framework: a case study. Clin Linguist Phon. 2015 Jan;29(1):59-75. doi: 10.3109/02699206.2014.956232. Epub 2014 Sep 12. PMID 25216375
- [Background] Benway NR, Preston JL, Hitchcock E, Rose Y, Salekin A, Liang W, McAllister T. Reproducible Speech Research With the Artificial Intelligence-Ready PERCEPT Corpora. J Speech Lang Hear Res. 2023 Jun 20;66(6):1986-2009. doi: 10.1044/2023_JSLHR-22-00343. Epub 2023 Jun 15. PMID 37319018